CLINICAL TRIAL: NCT04546373
Title: A Retrospective, Multicenter Study of Niraparib as Maintenance Therapy in Patients With Platinum Sensitive Recurrent Ovarian Cancer Who Have Received Niraparib Within the Expanded Access Program (EAP) in Spain
Brief Title: Niraparib as Maintenance Therapy in Patients With Platinum Sensitive Recurrent Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Responsible Party: Sponsor
Other Study IDs: GEICO 88-R
Record Dates: First submitted 2020-09-02; First posted 2020-09-14 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — niraparib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Niraparib — Patient's medical records will be screened by local clinical staff to assess for eligibility according to selection criteria. The study comprises a single study visit, in which the patient will give her informed consent to participate (when the patient is alive) and the physician will extract the study data from the patient's medical charts. All eligible deceased and consenting living patients at the participating centers will be included. Data will be directly retrieved from hospital medical records and reported in the electronic Case Report Form (eCRF).

SUMMARY:
In April 2017, Tesaro, Inc. opened an expanded access program (EAP) to make niraparib, an investigational poly (ADP-ribose) polymerase (PARP) inhibitor, available to eligible women with recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer following a complete or partial response to platinum-based chemotherapy, mainly for BRCA wild-type (BRCAwt) tumor patients, a clear unmet medical need for these ovarian cancer patients. As of 19 August 2019, the EAP closing date, there were 446 patients enrolled in 105 Spanish sites.

All eligible deceased and consenting living patients at the participating centers will be included. Data will be directly retrieved from hospital medical records and reported in the electronic Case Report Form (eCRF).

This study seeks to evaluate the safety profile and dose adjustments of niraparib in platinum sensitive recurrent ovarian cancer patients treated in a real world setting within the Spanish expanded access program (EAP).

ELIGIBILITY:
Inclusion Criteria:

* Female participants 18 years old or older.
* Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent.
* Participant must have received niraparib within the Spanish expanded access program (EAP).
* Patients must have received at least 1 week of treatment with niraparib.
* Histological diagnosis of high grade serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
* Participants must have completed at least 2 previous courses of platinum-containing therapy (e.g., carboplatin, oxaliplatin, or cisplatin).
* For the penultimate (next to last) platinum-based chemotherapy course prior to enrolment on the program the patient must have platinum sensitive disease after this treatment; defined as achieving a response (complete response (CR) or partial response (PR)) and disease progression occurring no sooner than 6 months, after completion of the last dose of platinum chemotherapy.
* For the last chemotherapy course prior to inclusion in the program the patient must have received a platinum-containing regimen for a minimum of 4 cycles.
* For the last chemotherapy course prior to inclusion in the program the Patient must have achieved a partial (PR) or complete (CR) tumor response.
* The last platinum regimen does not necessarily have to immediately follow the next to last (penultimate) platinum regimen. For example, if a patient received a non-platinum regimen between the penultimate platinum regimen and last platinum regimen, they could be eligible, so long as they meet all entry criteria.
* When entering the EAP, patients must have met the following:

  * Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
  * Adequate organ function - Absolute neutrophil count (ANC) ≥ (greater than or equal to) 1,500/μL.
  * Adequate organ function - Platelets ≥ (greater than or equal to) 100,000/μL.
  * Adequate organ function - Hemoglobin ≥ (greater than or equal to) 9 g/dL.
  * No transfusions of erythrocytes or platelets within 2 weeks prior to assessing adequate hematological blood counts as listed above.

Exclusion Criteria:

* Patients without medical record available (lost, empty or unretrievable clinical information).
* Patients who decline consent.
* Patients who are deceased with prior express order to preserve their data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with diagnosis of high grade serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer, with recurrent disease sensitive to platinum, treated within the Spanish niraparib EAP.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Demographics | Month 4-6
Medical History | Month 4-6
Ovarian Cancer Diagnosis | Month 4-6
Ovarian Cancer Treatments (pre-Niraparib) | Month 4-6
Baseline (pre-Niraparib) | Month 4-6
Niraparib Treatment | Month 4-6
Niraparib Disease Progression | Month 4-6
Best Response Assessment | Month 4-6
Niraparib-Related Adverse Events | Month 4-6
Relevant Concomitant Medications | Month 4-6
Death | Month 4-6
Survival Status | Month 4-6
Subsequent Therapies for Ovarian Cancer | Month 4-6

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Cueva Bañuelos, Dr., Principal Investigator — Complejo Hospitalario Universitario de Santiago de Compostela
Locations (57):
- Spain (57):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital Universari Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncología Badalona, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Institut Català d´ Oncologia-Hospital Duran y Reynals, L'Hospitalet de Llobregat, Barcelona
  - Consorci Sanitari de Terrassa, Rubí, Barcelona
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital Universitario de Galdakao, Galdakao, Bizkaia
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital Universitario de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Universitario Donostia, San Sebastián, Gipuzkoa
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Lluís Alcanyís de Xàtiva, Xàtiva, Valencia
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña (Juan Canalejo), A Coruña
  - Hospital Universitari Sant Joan d'Alacant, Alicante
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital del Mar, Barcelona
  - Clínica Corachan, Barcelona
  - Hospital Universitari Dexeus - Grupo Quirónsalud, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital General San Jorge, Huesca
  - Complejo Hospitalario de Jaén - Hospital Médico-Quirúrgico, Jaén
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario de La Princesa, Madrid
  - Clínica Universidad de Navarra, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Complejo Hospitalario Universitario de Pontevedra (Hospital Montecelo), Pontevedra
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario de Valme, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Cueva JF, Palacio I, Churruca C, Herrero A, Pardo B, Constenla M, Santaballa A, Manso L, Estevez P, Maximiano C, Legeren M, Marquina G, de Juan A, Quindos M, Sanchez L, Barquin A, Fernandez I, Martin C, Juarez A, Martin T, Garcia Y, Yubero A, Gallego A, Martinez Bueno A, Guerra E, Gonzalez-Martin A. Real-world safety and effectiveness of maintenance niraparib for platinum-sensitive recurrent ovarian cancer: A GEICO retrospective observational study within the Spanish expanded-access programme. Eur J Cancer. 2023 Mar;182:3-14. doi: 10.1016/j.ejca.2022.12.023. Epub 2022 Dec 29. PMID 36706655